CLINICAL TRIAL: NCT00589030
Title: A Treatment of Unresectable Hepatocellular Carcinoma With TheraSphere (Yttrium-90 Glass Microspheres): A HDE Treatment Use Protocol
Brief Title: Yttrium Y 90 Radiolabeled Glass Beads in Treating Patients With Liver Cancer That Cannot Be Removed by Surgery
Status: No longer available | Type: Expanded Access
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 06057; CHNMC-06057; CDR0000579146 (Registry Identifier: NCI PDQ); NCI-2010-00429 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-01-03; First posted 2008-01-09 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; advanced adult primary liver cancer; localized unresectable adult primary liver cancer; recurrent adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Brachytherapy

INTERVENTIONS:
Radiation: brachytherapy — The target dose of TheraSphere® is 80-150Gy
Radiation: yttrium Y 90 glass microspheres — The target dose of TheraSphere® is 80-150Gy

SUMMARY:
RATIONALE: Internal radiation therapy uses radioactive material placed directly into or near a tumor to kill tumor cells. Using radiolabeled glass beads to kill tumor cells may be effective treatment for liver cancer that cannot be removed by surgery.

PURPOSE: To provide expanded access and study the side effects of yttrium Y 90 glass microspheres in treating patients with liver cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Provide supervised access to treatment with yttrium Y 90 glass microspheres (TheraSphere®) to eligible patients with primary cancer to the liver and who are not surgical resection candidates.
* Evaluate patient experience and toxicities associated with TheraSphere® treatment.
* Enter treatment experience into a liver database.

Secondary

* Determine the tumor response rates in patients receiving this treatment.

OUTLINE: This is a humanitarian device exemption use study.

Patients receive yttrium Y 90 glass microspheres (TheraSphere®) via percutaneous hepatic arterial infusion. Patients may be retreated between 30-90 days after the initial infusion.

After completion of study therapy, patients are followed for 30 days and then annually thereafter for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of hepatocellular carcinoma
* Surgical evaluation by a member of the Liver Tumor Program must conclude the patient is not a candidate for resection or ablation
* Eastern Cooperative Oncology Group (ECOG) Performance Status Score 0-2
* Able to comprehend and provide written informed consent in accordance with institutional and federal guidelines

Exclusion Criteria:

* Absolute granulocyte count =<1,500/ul
* Platelet count =<75,000/ul
* Serum creatinine >= 2.0 mg/dl
* Serum bilirubin

  * >= 2.0 mg/dl for bilateral treatment or lobar treatment
  * >= 3.0 mg/dl for single lesion which could be treated by segmental fusion
* History of severe allergy or intolerance to any contrast media, narcotics, sedatives, or atropine
* Bleeding, diathesis not correctable by usual forms of therapy
* Severe peripheral vascular disease that would preclude catheterization
* Portal hypertension with portal venous shunt away from the liver
* Evidence of potential delivery greater than 16.5 mCi (30 Gy absorbed dose) of radiation to the lungs on either:

  1. first TheraSphere administration; or
  2. cumulative delivery of radiation to the lungs > 30 Gy over multiple treatments
* Evidence of any detectable Tc-99m MMA flow to the stomach or duodenum, after application of established angiographic techniques to stop such flow
* Significant extrahepatic disease representing an imminent life-threatening outcome
* Severe liver dysfunction (Childs' Classification C) or pulmonary insufficiency (requiring continuous oxygen therapy)
* Active uncontrolled infection
* Significant underlying medical or psychiatric illness
* Pregnant women may not participate
* Children may not participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Jen Chen, MD, PhD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States